CLINICAL TRIAL: NCT04283292
Title: Capsaicin for the Treatment of Cannabinoid Hyperemesis Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Angela Holian, Emergency Medicine Clinical Pharmacist, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21957
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2021-01

CONDITIONS: Cannabinoid Hyperemesis Syndrome
MeSH Terms: conditions — Cannabinoid Hyperemesis Syndrome | interventions — Capsaicin

STUDY DESIGN:
Intervention Model Description: Randomized to capsaicin or placebo in a 1:1 ratio (like the flip of a coin).
Who Masked: Care Provider, Investigator
Masking Description: investigational pharmacists and designated personell will the only unblinded study staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Capsaicin (Experimental): capsaicin 0.075% cream applied once topically
  Interventions: Drug: Capsaicin
- Placebo (Active Comparator): placebo cream applied once topically
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Capsaicin — Topical Capsaicin for the treatment of Cannabinoid Hyperemesis Syndrome
  Other Names: Zostrix
  Arms: Capsaicin
Drug: Placebo — Placebo cream that is applied once topically
  Arms: Placebo

SUMMARY:
This study aims to determine if capsaicin cream offers symptomatic relief to patients suffering from Cannabinoid Hyperemesis Syndrome (condition that leads to repeated and severe bouts of vomiting).

DETAILED DESCRIPTION:
Objectives:

The purpose of this study is to determine if capsaicin cream offers symptomatic relief to patients suffering from Cannabinoid Hyperemesis Syndrome. We hypothesize that the use of topical capsaicin may provide effective symptomatic relief more quickly than conventional anti-emetic therapy alone thereby decreasing costs for continued drug therapies, repeat laboratory testing, radiographic imaging, and specialist consults.

Primary endpoint:

Time to resolution of symptoms, clinical improvement in pain score as defined by visual analog score.

Approach and methods:

Patients presenting to the UVA Emergency Department with chief complaint of nausea and vomiting who endorse cannabinoid use via inhalation or consumption. Patients 18 years of age and older will be included in the study and patients who have another clear indication for nausea/vomiting or cyclic vomiting (infection, appendicitis, pain, etc.) will be excluded. Patients who are enrolled in the study will be randomized 1:1 to treatment vs. placebo. All patients will be allowed 1L of intravenous fluids and one to two standard anti-emetics. The Investigational Drug Services team at UVA will be involved in compounding the capsaicin treatment versus placebo and drug/placebo shall remain in place for at least 30 minutes. Clinical improvement will be scored based on visual analog score for pain and assessment at hourly increments until discharge or admission.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Diagnosis of cannabinoid hyperemesis syndrome

Exclusion Criteria:

* Patients who receive more than 2 anti-emetic therapies prior to screening for enrollment
* Patients who receive haloperidol as an anti-emetic therapy
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Time to resolution of symptoms | 1 day (During emergency department admission)
  Time that it takes for symptoms to be resolved for those with Cannabinoid Hyperemesis Syndrome

SECONDARY OUTCOMES:
Clinical improvement in pain score | 1 day (During emergency department admission)
  Clinical improvement in pain score as defined by visual analog score with a scale from 0-10 where is 0 is no pain and 10 is unbearable pain. Pain should decrease over time and this will be measure by the visual analog scale

OTHER OUTCOMES:
Symptom improvement at thirty days | 30 days (outpatient phone call)
  Follow-up phone call at thirty days to investigate any symptom improvement or change in cannabinoid usage.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Holian, PharmD, Principal Investigator — University of Virginia
Locations (1):
- UVA Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No